CLINICAL TRIAL: NCT05389371
Title: Use of a Virtual Weight Management Program to Enable Weight Loss and Improve Metabolic Health and Quality of Life for Patients With Osteoarthritis and Obesity
Brief Title: OA Optimization Program Pilot Trial
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Calgary (Other)
Collaborators: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: REB19-1814
Record Dates: First submitted 2022-05-19; First posted 2022-05-25 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2023-11

CONDITIONS: Osteo Arthritis Knee; Osteoarthritis, Knee; Osteoarthritis, Hip; Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis, Hip; Osteoarthritis | interventions — Physical Therapy Modalities; Educational Status; Exercise

STUDY DESIGN:
Intervention Model Description: parallel-arm randomized trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alberta Healthy Living Program (Active Comparator): An integrated community-based chronic disease management program available to residents of Alberta.
  Interventions: Behavioral: Alberta Healthy Living Program; Behavioral: Osteoarthritis advice; Behavioral: Physiotherapy
- Alberta Obesity Centre Program (Experimental): Evidence-based medical management of obesity using a multidisciplinary approach.
  Interventions: Behavioral: Alberta Obesity Centre Program; Behavioral: Osteoarthritis advice; Behavioral: Physiotherapy

INTERVENTIONS:
Behavioral: Alberta Healthy Living Program — Weight management services
  Arms: Alberta Healthy Living Program
Behavioral: Alberta Obesity Centre Program — Multi-disciplinary obesity management
  Arms: Alberta Obesity Centre Program
Behavioral: Osteoarthritis advice — Living Your Best Life with Osteoarthritis Handbook
Behavioral: Physiotherapy — GLA:D physiotherapy programs.
  Other Names: GLA:D (TM) education and exercise

SUMMARY:
Total joint replacement is a highly successful treatment option for people affected by severe osteoarthritis (OA), however, the mismatch between resources and demand for this surgery means that many patients face long wait times while enduring worsening pain and disability. The Alberta Hip and Knee Program is a centralized intake system for patients referred for total joint replacement assessment. Over 3000 patients are assessed annually at the Calgary location (Alberta Hip and Knee Clinic at Gulf Canada Square) where previously patients waited an average of 43 weeks for a surgical consult then an additional 30 weeks until surgery. Given that many elective surgeries in Alberta have been cancelled in response to the COVID19 pandemic, these wait times have increased significantly, with no clearing of the surgical backlog for the foreseeable future. Long wait times for patients can become a spiral of more debility, less mobility, and subsequent weight gain. The current standard of care for patients with obesity awaiting surgery provides little support or guidance beyond general advice about the importance of a healthy weight and remaining active. This waiting period represents an untapped window of opportunity to intervene and help patients with obesity and OA to lessen their disease burden and improve overall health, while addressing patient priorities such as regaining lost function and improving quality of life.

Many patients with osteoarthritis also have obesity. The best practices in obesity treatment requires a multidisciplinary approach. Our aim is to conduct a pilot randomized controlled trial (RCT) to evaluate the feasibility of incorporating the multidisciplinary Alberta Obesity Centre program into the clinical care pathway for patients with obesity and OA while they await surgical evaluation at the Alberta Hip and Knee Clinic at Gulf Canada Square. The results of this feasibility trial will help inform a larger scale trial that will be powered for clinical and health economics outcomes.

ELIGIBILITY:
Inclusion Criteria:

* body mass index (weight in kilograms divided by height in metres squared) greater than 30
* symptomatic osteoarthritis (referred to the Alberta Hip and Knee Clinic for assessment for total joint replacement surgery)

Exclusion Criteria:

* Currently following a specialized or therapeutic diet
* pregnant or breastfeeding
* diagnosed with type 1 diabetes
* unable to read or speak English
* unable to use email
* unable to use virtual platforms such as Zoom

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-06-28 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Determine the number of adults with osteoarthritis and obesity that are eligible to participate in the trial | 0-12 months
  The number of patients approached
The number of these adults with osteoarthritis and obesity who would be willing to take part in this trial | 0-12 months
  The number of patients who actually enroll
The characteristics of these adults with osteoarthritis and obesity who are willing to take part in the trial | 0-12 months
  Patient sex, gender, age, and medical history
The number and percentage of participants retained at 12-months | 0-12 months
  Number and percentage of patients attending at 12-month follow up and reasons for drop-out

SECONDARY OUTCOMES:
Change in body mass | 0-12 months
  Change in body mass (weight loss)
Decision to proceed with joint replacement surgery | 12 months
  Yes/no decision to proceed with joint replacement surgery
Change in waist circumference | 0-12 months
  waist circumference (centimetres)
Change in blood pressure | 0-12 months
  blood pressure (millimetres of mercury)
Change in blood lipid profile | 0-12 months
  blood lipids
Change in glycemic control | 0-12 months
  glycated hemoglobin (HbA1c)
Change in quality of life | 0-12 months
  Quality of life measured by the Alberta Bone and Joint Health Institute Hip and Knee Replacement Outcomes Tool
Change in medication usage | 0-12 months
  All prescription medications will be tracked and recorded by a study physician

CONTACTS AND LOCATIONS:
Locations (1):
- University of Calgary, Calgary, Alberta, Canada